CLINICAL TRIAL: NCT05593211
Title: Feasibility Study of the Kronos Electrocautery Device
Brief Title: Assess Safety and Performance of the Kronos Electrocautery Device for Electrocautery Procedures Following Coaxial Biopsy Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Single Pass Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SP-01
Record Dates: First submitted 2022-08-19; First posted 2022-10-25 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Hepatic Disease; Renal Disease
Keywords: Hepatitis; Liver Disease; Hepatic Disease
MeSH Terms: conditions — Digestive System Diseases; Kidney Diseases; Hepatitis; Liver Diseases

STUDY DESIGN:
Intervention Model Description: The Kronos Electrocautery Device is a disposable electrocautery device that can cauterize deep tissue through a standard biopsy procedure guide needle. This device is intended to coagulate the tissue surrounding the core biopsy channel during withdrawal to reduce or eliminate significant post-procedural bleeding. Currently, the Kronos Electrocautery Device consists of one (1) size. As such, the existing Kronos Electrocautery Device is chosen as the worst-case condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Patients undergoing a scheduled, elective, solid organ biopsy procedures on the liver or kidneys (Experimental)
  Interventions: Device: Kronos Electrocautery Device

INTERVENTIONS:
Device: Kronos Electrocautery Device — The Kronos Electrocautery Device is a disposable electrocautery device that can cauterize deep tissue through a standard biopsy procedure guide needle. This device is intended to coagulate the tissue surrounding the core biopsy channel during withdrawal to reduce or eliminate significant post-procedural bleeding. Currently, the Kronos Electrocautery Device consists of one (1) size. As such, the existing Kronos Electrocautery Device is chosen as the worst-case condition

SUMMARY:
The primary objective for this study is to assess safety and performance of the Kronos Electrocautery Device for electrocautery procedures following coaxial biopsy procedures on areas that include, but are not limited to, liver, kidney, lungs, breasts, soft tissue, etc.

DETAILED DESCRIPTION:
The Kronos Electrocautery Device is intended to be used in electrocautery procedures to control bleeding by use of electrical current to heat the device probe tip that is applied directly to the target tissue area of treatment. Prospective, multi-center, single-arm study with consecutive, eligible subject enrollment at each site. Patients who require a coaxial biopsy procedures on areas that include, but are not limited to, liver, kidney, lungs, breasts, soft tissue, etc., will be eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing a scheduled, elective, coaxial biopsy procedures on areas that include, but are not limited to, liver, kidney, lungs, breasts, soft tissue, etc.,
2. Patients have signed an informed consent
3. Patients who are ≥ 18 years of age

Exclusion Criteria:

1. Patients with known bleeding disorder
2. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
3. Women of childbearing potential who are pregnant, lactating, or planning to become pregnant during the course of the clinical investigation.
4. Active illness or active systemic infection or sepsis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Tahour, MD, Principal Investigator — Long Beach Memorial Medical Center
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whittier WL, Korbet SM. Timing of complications in percutaneous renal biopsy. J Am Soc Nephrol. 2004 Jan;15(1):142-7. doi: 10.1097/01.asn.0000102472.37947.14. PMID 14694166
- [Background] Manno C, Strippoli GF, Arnesano L, Bonifati C, Campobasso N, Gesualdo L, Schena FP. Predictors of bleeding complications in percutaneous ultrasound-guided renal biopsy. Kidney Int. 2004 Oct;66(4):1570-7. doi: 10.1111/j.1523-1755.2004.00922.x. PMID 15458453
- [Background] Mahal AS, Knauer CM, Gregory PB. Bleeding after liver biopsy. West J Med. 1981 Jan;134(1):11-4. PMID 7210659
- [Background] Lim S, Rhim H, Lee MW, Song KD, Kang TW, Kim YS, Lim HK. New Radiofrequency Device to Reduce Bleeding after Core Needle Biopsy: Experimental Study in a Porcine Liver Model. Korean J Radiol. 2017 Jan-Feb;18(1):173-179. doi: 10.3348/kjr.2017.18.1.173. Epub 2017 Jan 5. PMID 28096727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Undergoing a Scheduled, Elective, Solid Organ Biopsy Procedures on the Liver or Kidneys
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing a Scheduled, Elective, Solid Organ Biopsy Procedures on the Liver or Kidneys
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Absence of Hematoma Formation
Description: Patients will be contacted on day 14 post-procedure and asked a series of questions regarding Adverse Events related to the procedure.
Time Frame: 14 days
Population: The patients that completed the study.
Measure: Number; unit: participants
Arm/Group | Patients Undergoing a Scheduled, Elective, Solid Organ Biopsy Procedures on the Liver or Kidneys
Number analyzed (Participants) | 30
participants | 30

2. Primary Outcome: Measure and Categorize Amount of Blood Loss From Biopsy Access Site
Description: The weight of 10 gauze pads is taken prior to the procedure. Post-procedure, those same 10 gauze pads used at biopsy access site are weighed again to measure in grams, the amount of blood loss. The scale ranges from 1 (unacceptable) to 5 (excellent).
Time Frame: 1 hour post procedure
Population: Number of patients that completed the study
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients Undergoing a Scheduled, Elective, Solid Organ Biopsy Procedures on the Liver or Kidneys
Number analyzed (Participants) | 30
score on a scale | 5.0 [1 to 5]

3. Primary Outcome: Absence of the Need for Ultrasound Examination Due to Observation of Bleeding
Description: Measuring the amount of patient who did not need an ultrasound examination due to observation of bleeding
Time Frame: 8 hours post procedure
Population: amount of patients completed the study
Measure: Number; unit: participants
Arm/Group | Patients Undergoing a Scheduled, Elective, Solid Organ Biopsy Procedures on the Liver or Kidneys
Number analyzed (Participants) | 30
participants | 30

4. Secondary Outcome: Absence of Secondary Reintervention
Description: Patients will be contacted on day 14 post-procedure and asked a series of questions regarding Adverse Events related to the procedure. Measuing the amount of patients who did not require secondary reintervention.
Time Frame: 14 days
Population: 30 patients that completed the study
Measure: Number; unit: participants
Arm/Group | Patients Undergoing a Scheduled, Elective, Solid Organ Biopsy Procedures on the Liver or Kidneys
Number analyzed (Participants) | 30
participants | 30

5. Secondary Outcome: Time to Hospital Discharge
Time Frame: 8 hours post procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 days post proceedure
Arm/Group | Patients Undergoing a Scheduled, Elective, Solid Organ Biopsy Procedures on the Liver or Kidneys
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Undergoing a Scheduled, Elective, Solid Organ Biopsy Procedures on the Liver or Kidneys (N=30)
Trace Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Trace pneumothorax (right side) following biopsy & Kronos single pass use. Not characterized as procedure or device-related. Mild severity.
Shortness of breath and coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Notified at 14-day followup. Worsening shortness of breath after biopsy and coughing up pink sputum. Not characterized as procedure or device-related. Mild severity. No intervention was necessary.
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Notified at 14-day follow-up. Not characterized as device-related. Moderate severity. Pre-existing condition.
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Notified at 14-day follow-up. Not characterized as device-related. Mild severity. Pain was present before biopsy due to metastatic disease of numerous organs.
Anasarca (Skin and subcutaneous tissue disorders) | 1 (1) — Notified at 14-day follow-up. Not characterized as device-related. Mild severity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT05593211/Prot_SAP_000.pdf